CLINICAL TRIAL: NCT07108595
Title: Efficacy and Safety of T-DXd in Patients With HER2-positive and HER2-low Metastatic Breast Cancer: a Real-world Study
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20250729TDXd
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: HER2-positive; HER2-low; T-DXd; Real-world study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Patients receive T-DXd
  Interventions: Drug: T- Dxd

INTERVENTIONS:
Drug: T- Dxd — T-DXd based therapy

SUMMARY:
Evaluate the efficacy and safety of T-DXd in patients with HER2-positive and HER2-low metastatic breast cancer

DETAILED DESCRIPTION:
The DESTINY-Breast trials established trastuzumab deruxtecan (T-DXd) as a treatment significantly improving outcomes in human epidermal growth factor receptor 2 (HER2)-positive and HER2-low metastatic breast cancer (MBC). However, real-world effectiveness is susceptible to confounding factors. This multicenter, real-world study aims to systematically evaluate the efficacy and safety of T-DXd in patients with HER2-positive and HER2-low MBC. Key clinicopathological parameters were to be integrated to develop an individualized prognostic prediction model, facilitating precision medicine implementation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. female patients aged ≥18 years;
2. histologically confirmed HER2-positive (IHC 3+ or IHC 2+/FISH+) or HER2-low (IHC 1+ or IHC 2+/FISH-) disease;
3. radiologically confirmed recurrent or metastatic disease;
4. completion of ≥2 cycles of T-DXd therapy;
5. comprehensive medical documentation;
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤3;
7. measurable target lesions according to RECIST 1.1

Exclusion Criteria:

1. history of interstitial lung disease
2. incomplete medical records
3. concurrent malignancies;
4. pregnancy or lactation
5. psychiatric disorders compromising treatment adherence

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive or HER2-low expressing, locally advanced or metastatic breast cancer were eligible and received therapy. DXd was administered intravenously at 5.4 mg/kg every 3 weeks (21-day cycles) until disease progression or unacceptable toxicity. Dose adjustments were performed according to clinical status and treatment tolerance. Complete blood count with hepatic and renal function parameters were monitored before each cycle. Tumor response assessment via RECIST 1.1 criteria was conducted radiologically every two cycles.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Adverse Events (AE) | 2 years
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, JiangSu 210000, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No